CLINICAL TRIAL: NCT01329367
Title: Efecto de Una Intervención Dietética Sobre La Expresión De Genes De La Inflamación Y El Estrés Oxidativo En Niños Obesos
Brief Title: Nutrigenomics And Children Obesity: A Moderate Weight Loss Intervention Study
Acronym: NUGENOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hospital Virgen del Camino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUGENOI-UN
Record Dates: First submitted 2011-01-20; First posted 2011-04-05 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: EVASYON; GENOI; antioxidants; legume; fish
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Control group: Subjects will receive Nutritional education together with weight management counselling for overweight and obesity.
  -10 weekly personal interviews with a registered nutritionist for body weight control.
  Interventions: Behavioral: Control group
- Protein group (Experimental): Protein group: Participants will receive Nutritional education and personalised structured meal plan with a calorie restricted diet (20-40% of the subject's energy expenditure at baseline) according to obesity degree, encouraging high consumption of legumes and fish (protein rich diets).
  -10 weekly personal interviews with a registered nutritionist for body weight control.
  Interventions: Behavioral: Protein group
- Antioxidant group (Experimental): Antioxidant group: Participants will receive Nutritional education and personalized structured meal plan with a calorie restricted diet (20-40% of the subject's energy expenditure at baseline) according to obesity degree, encouraging high consumption of fruits and vegetables (antioxidant rich diets).
  -10 weekly personal interviews with a registered nutritionist for body weight control.
  Interventions: Behavioral: Antioxidant group

INTERVENTIONS:
Behavioral: Control group — Subjects will receive Nutritional education together with weight management counselling for overweight and obesity.
  -10 weekly personal interviews with a registered nutritionist for body weight control.
  Arms: Control group
Behavioral: Protein group — Participants will receive Nutritional education and personalised structured meal plan with a calorie restricted diet (20-40% of the subject's energy expenditure at baseline) according to obesity degree, encouraging high consumption of legumes and fish (protein rich diets).
  -10 weekly personal interviews with a registered nutritionist for body weight control.
  Arms: Protein group
Behavioral: Antioxidant group — Participants will receive Nutritional education and personalized structured meal plan with a calorie restricted diet (20-40% of the subject's energy expenditure at baseline) according to obesity degree, encouraging high consumption of fruits and vegetables (antioxidant rich diets).
  -10 weekly personal interviews with a registered nutritionist for body weight control.
  Arms: Antioxidant group

SUMMARY:
The consumption of diets enriched in proteins (legumes and fish) or antioxidant (fruits and vegetables) could have beneficial effects beyond those of the caloric restriction on biomarkers of the inflammatory and oxidative status. OBJECTIVE: To address the effect of a 10-week dietary intervention aimed to weight loss in obese or overweight children (7-15 aged) on genomics, particularly the changes in the expression of genes related to the inflammatory status and oxidative stress. METHODOLOGY: 44 Navarra children and adolescents of both sexes from Pediatric Endocrinology Services at different Hospitals in Pamplona will be recruited. The effect of the intensive consumption of different groups of food will be evaluated: legumes and fish ( diets in proteins) and vegetable and fruits (rich diets in antioxidants). Before and after the intervention, the following items will be analyzed: (1) the diet of the subjects, (2) body composition and 3 magnitudes related to biological and development parameters, being: (3) lipid and metabolic phenotypic profile; (4) markers of the inflammatory status and oxidative stress, and (5) the genomic profile. The dietary programme will be implemented both in group workshops addresseded to patients and their family, and in individual sessions with the pediatricians and/or registered dieticians. Finally, the programme efficacy will be evaluated by the scoreboards integrated in the 5 variables already mentioned.

DETAILED DESCRIPTION:
A longitudinal intervention study in 44 overweight and obese adolescents (23 females and 21 males; mean age 11.5 years) for 10 weeks based on a calorie restricted diet (20-40%) according to obesity degree.

ELIGIBILITY:
Inclusion Criteria:

* Children between 7 and 15 years
* Body Mass Index (BMI) higher to 97 percentile. (Cole et al, 2000)*

  * Cole TJ, Belizzy MC, Flegal KM, Dietz WH. Br Med J 2000; 320: 1-6.

Exclusion Criteria:

* Use of prescription medication
* To suffer from any major psychiatry or neurological disease, bulimia nervosa, familiar hypercholesterolemia or any major cardiac, or respiratory metabolic disease.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Body masss index | week 0
  Body mas index will be measured at the beginning of the study (week 0), at week 5 and week 10 (end of the study).

SECONDARY OUTCOMES:
Basal glucose concentration | week 10
  Basal glucose concentration will be measured at the beginning of the study (week 0)and week 10 (end of the study).
Insulin concentrations | week 0
  Insulin concentrations will be analysed at week 0, and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Marti, PhD, BPharm, Principal Investigator — University of Navarra; Cristina Azcona, MD, Study Director — University of Navarre Clinic; Maria Chueca, MD, Study Chair — Virgen del Camino Hospital
Locations (2):
- Spain (2):
  - UNavarre, Pamplona, Navarre
  - University of Navarre, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rendo-Urteaga T, Garcia-Calzon S, Gonzalez-Muniesa P, Milagro FI, Chueca M, Oyarzabal M, Azcona-Sanjulian MC, Martinez JA, Marti A. Peripheral blood mononuclear cell gene expression profile in obese boys who followed a moderate energy-restricted diet: differences between high and low responders at baseline and after the intervention. Br J Nutr. 2015 Jan 28;113(2):331-42. doi: 10.1017/S0007114514003584. Epub 2014 Dec 4. PMID 25471305
- [Result] Rendo-Urteaga T, Puchau B, Chueca M, Oyarzabal M, Azcona-Sanjulian MC, Martinez JA, Marti A. Total antioxidant capacity and oxidative stress after a 10-week dietary intervention program in obese children. Eur J Pediatr. 2014 May;173(5):609-16. doi: 10.1007/s00431-013-2229-7. Epub 2013 Dec 6. PMID 24310523
- [Result] Rendo-Urteaga T, Garcia-Calzon S, Martinez-Anso E, Chueca M, Oyarzabal M, Azcona-Sanjulian MC, Bustos M, Moreno-Aliaga MJ, Martinez JA, Marti A. Decreased cardiotrophin-1 levels are associated with a lower risk of developing the metabolic syndrome in overweight/obese children after a weight loss program. Metabolism. 2013 Oct;62(10):1429-36. doi: 10.1016/j.metabol.2013.05.011. Epub 2013 Jul 12. PMID 23856329
- [Result] Ojeda-Rodriguez A, Morell-Azanza L, Azcona-Sanjulian MC, Martinez JA, Ramirez MJ, Marti A. Reduced serotonin levels after a lifestyle intervention in obese children: association with glucose and anthropometric measurements. Nutr Hosp. 2018 Mar 1;35(2):279-285. doi: 10.20960/nh.1439. PMID 29756959
- [Result] Morell-Azanza L, Garcia-Calzon S, Rendo-Urteaga T, Martin-Calvo N, Chueca M, Martinez JA, Azcona-Sanjulian MC, Marti A. Serum oxidized low-density lipoprotein levels are related to cardiometabolic risk and decreased after a weight loss treatment in obese children and adolescents. Pediatr Diabetes. 2017 Aug;18(5):392-398. doi: 10.1111/pedi.12405. Epub 2016 Jul 20. PMID 27435258
- [Result] Marti A, Morell-Azanza L, Rendo-Urteaga T, Garcia-Calzon S, Ojeda-Rodriguez A, Martin-Calvo N, Moreno-Aliaga MJ, Martinez JA, Azcona-San Julian MC. Serum and gene expression levels of CT-1, IL-6, and TNF-alpha after a lifestyle intervention in obese children. Pediatr Diabetes. 2018 Mar;19(2):217-222. doi: 10.1111/pedi.12561. Epub 2017 Jul 27. PMID 28749076